CLINICAL TRIAL: NCT05407376
Title: Produce Prescriptions At Kaiser Permanente Southern California - an Innovative 'food As Medicine' Clinical Trial to Improve Food Insecurity and Health Among Medicaid Patients with Consistently Uncontrolled Type 2 Diabetes
Brief Title: Food As Medicine Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12876
Record Dates: First submitted 2022-04-08; First posted 2022-06-07 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention- High Dose (Active Comparator): Participation will last approximately 6 months. Participants enrolled in the high-dose intervention arm will receive a weekly produce delivery directly to their home in addition to the completion of 3 questionnaires and collection of the HbA1c at the end of study.
  Interventions: Other: Produce prescription (weekly produce delivery)
- Intervention-Low Dose (Active Comparator): Participation will last approximately 6 months. Participants enrolled in the low-dose intervention arm will receive a weekly produce delivery directly to their home in addition to the completion of 3 questionnaires and collection of the HbA1c at the end of study. The amount of produce provided in this arm will be lower per month per household size than the high dose arm.
  Interventions: Other: Produce prescription (weekly produce delivery)
- Usual Care (No Intervention): Participation will last approximately 6 months. Participants enrolled in the Usual Care arm will complete 3 questionnaires and collection of the HbA1c at the end of study.

INTERVENTIONS:
Other: Produce prescription (weekly produce delivery) — Participants will receive weekly produce deliveries and recipes sent directly to their homes for 6 months.
  Arms: Intervention- High Dose; Intervention-Low Dose

SUMMARY:
The investigators are conducting a pre-randomized controlled trial to assess the effect of a 6 month Produce Prescription intervention for patients enrolled in Medicaid who experience consistently uncontrolled Hemoglobin A1c (HbA1c). The study is conducted at Kaiser Permanente Southern California, a large and diverse integrated health care system that serves 4.7 million members. Eligible participants are members aged 18 or older, currently enrolled in Medicaid who were diagnosed with diabetes for at least 24 months and had at least two Hba1c measurements of 7.5% or higher in the past 12 months. Patients in the intervention arm may enroll in tele nutrition counseling. The study team will recruit a total of 450. Participants, will be pre-randomized into one of three arms, 1) high dose intervention arm, a 2) low dose intervention and 3) a usual care group to achieve 150 participants enrolled in each arm. Produce is delivered weekly for participants of both intervention arms. Participants randomized to the high dose arm will receive a greater amount per month of produce versus the low dose amount (for a family of 3-4, $180 per month versus $135 respectively). Foods are provided along with recipes. The amount of food delivered is adjusted for each additional family member for up to 5 family members. The primary outcome is change in hemoglobin A1c pre-intervention and 6 months after enrollment. Secondary outcomes include, food insecurity status, dietary intake and other patient reported outcomes related to barriers to healthy eating including family conflict and cooking habits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Diagnosed with Type 2 Diabetes for at least 24 months
* Diagnosed with Type 2 Diabetes and have at least two HbA1cs of 7.5% or higher in 12 months prior to recruitment
* Have MediCaid insurance at the time of their last hba1c test
* Will be able to provide informed consent
* Will be able to consent to research activities, including receiving a weekly produce box
* Will be able to receive and prepare delivered foods

Exclusion Criteria:

* Pregnant women
* Living in a board and care where your meals are provided for you
* Unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c between baseline and 6 months | Baseline and 6 months after baseline assessment
  Both intervention and control participants will have their HbA1c tested at baseline and 6 months after the baseline assessment.

SECONDARY OUTCOMES:
Analyze the difference in difference of patient-reported food security between the intervention and control group. | Survey completed at Baseline, 3 months and 6 months
  Calculated by the change in self-reported food security using the US Adult Food Security Short Form (a six-item self-administered patient survey to identify food-insecure households and households with very low food security). Scores range from 0 (high or marginal food security) to 6 (very low food security).
Analyze the difference in difference of patient-reported food-related self management between the intervention and control group. | Survey completed at Baseline, 3 months and 6 months
  Calculated by the change in self-reported food-related self management.
Analyze the difference in difference of patient-reported diet quality between the intervention and control group. | Survey completed at Baseline, 3 months and 6 months
  Calculated by the change in self-reported food security using an adapted Rapid Eating Assessment of Participants Short form survey (REAP-S), which is a tool used to help care providers quickly assess a participant's diet.
Analyze the difference in difference of patient-reported nutritional security between the intervention and control group. | Survey completed at Baseline, 3 months and 6 months
  Calculated by change in self-reported nutrition security.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia L Nau, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Southern California, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No